CLINICAL TRIAL: NCT07329829
Title: Comparison of Postoperative Analgesic Efficacy of Preoperative Pericapsular Nerve Group (PENG) Block With PENG Block and Lateral Femoral Cutaneous Nerve Block in Lateral Incision Hip Surgery
Brief Title: Perioperative Analgesic Effects of PENG Versus PENG Plus LFCN Block in Hip Surgeries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, ASSOCIATE PROFESSOR, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSH-ANES-MG-01
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-07

CONDITIONS: HİP FRACTURE; Hip Surgery (Lateral Incision); Postoperative Pain Management; Analgesia, Postoperative; Regional Anesthesia Success
Keywords: Pericapsular Nerve Group Block (PENG Block); Lateral Femoral Cutaneous Nerve Block (LFCN Block); Hip Surgery; Regional Anesthesia; Postoperative Analgesia; Pain Control; Opioid Consumption; Early Mobilization
MeSH Terms: conditions — Hip Fractures; Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG BLOCK GROUP (Experimental): An ultrasound-guided Pericapsular Nerve Group (PENG) block will be performed preoperatively using standard local anesthetic techniques to provide postoperative analgesia in patients undergoing lateral incision hip surgery.
  Interventions: Procedure: Pericapsular nerve group (PENG) block
- PENG + LFCN BLOCK GROUP (Experimental): Patients in this group will receive a preoperative ultrasound-guided Pericapsular Nerve Group (PENG) block combined with a Lateral Femoral Cutaneous Nerve (LFCN) block for postoperative analgesia prior to lateral incision hip surgery under spinal anesthesia.
  Interventions: Procedure: Pericapsular nerve group (PENG) block; Procedure: Lateral Femoral Cutaneous Nerve (LFCN) Block

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block — An ultrasound-guided Pericapsular Nerve Group (PENG) block will be performed preoperatively using standard local anesthetic techniques to provide postoperative analgesia in patients undergoing lateral incision hip surgery.
Procedure: Lateral Femoral Cutaneous Nerve (LFCN) Block — An ultrasound-guided Lateral Femoral Cutaneous Nerve (LFCN) block will be performed preoperatively as an adjunct to the PENG block to enhance postoperative analgesia in patients undergoing lateral incision hip surgery.
  Arms: PENG + LFCN BLOCK GROUP

SUMMARY:
This study is designed to find the best way to control pain after hip surgery performed through a side (lateral) incision. Two different types of nerve blocks used before the operation will be compared.

In one group, patients will receive a Pericapsular Nerve Group (PENG) block, which numbs the main nerves that carry pain signals from the hip joint. In the other group, patients will receive a PENG block together with a Lateral Femoral Cutaneous Nerve (LFCN) block, which adds extra pain relief for the skin and outer part of the thigh.

A total of 72 patients between 18 and 80 years old will take part in this study. All operations will be done under spinal anesthesia. Pain levels will be measured several times during the first 24 hours after surgery using a simple 0-10 pain scale. Patients will receive pain medicine through a pump that allows them to press a button when they feel pain. The total amount of medicine used will be recorded.

The researchers will also monitor when patients first need pain medicine, when they can start walking, how satisfied they are with pain control, and if they experience side effects such as nausea or dizziness.

By comparing the two methods, the study aims to see whether adding the LFCN block to the PENG block provides better pain control, lower drug use, faster recovery, and higher patient comfort after hip surgery.

DETAILED DESCRIPTION:
Postoperative pain following hip surgery remains a significant clinical challenge, particularly in procedures performed through a lateral incision, where both deep articular and superficial cutaneous pain components contribute to patient discomfort. Effective regional anesthesia techniques are essential to optimize postoperative analgesia, facilitate early mobilization, and reduce opioid-related adverse effects.

The Pericapsular Nerve Group (PENG) block has been introduced as a motor-sparing regional anesthesia technique targeting the articular branches of the femoral, obturator, and accessory obturator nerves, providing effective analgesia for hip joint-related pain. However, due to its limited coverage of cutaneous innervation, patients undergoing lateral incision hip surgery may continue to experience residual superficial pain.

The Lateral Femoral Cutaneous Nerve (LFCN) block selectively targets the sensory innervation of the anterolateral thigh and may complement the PENG block by addressing the cutaneous component of postoperative pain. The combined use of PENG and LFCN blocks has the potential to provide more comprehensive analgesia without compromising motor function.

This study is designed to evaluate whether the addition of an LFCN block to a standard PENG block enhances postoperative pain control and recovery outcomes in patients undergoing hip surgery via a lateral approach. By comparing these two regional anesthesia strategies, the study aims to contribute evidence-based guidance for optimizing multimodal analgesia protocols in hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years
* Patients scheduled for elective or trauma-related hip surgery performed through a lateral incision under spinal anesthesia
* Patients receiving a preoperative ultrasound-guided Pericapsular Nerve Group (PENG) block or a PENG block combined with a Lateral Femoral Cutaneous Nerve (LFCN) block
* American Society of Anesthesiologists (ASA) physical status I-III
* Patients with full orientation and the ability to cooperate
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Contraindications to regional anesthesia, including coagulopathy or local infection at the injection site
* Presence of neuropathic disorders or conditions that may affect pain perception, including chronic analgesic use
* Requirement for conversion to general anesthesia
* Postoperative admission to the intensive care unit
* Known allergy or hypersensitivity to opioids or local anesthetics
* American Society of Anesthesiologists (ASA) physical status IV-V

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (NRS Score) | 2, 6, 12, and 24 hours postoperatively
  Postoperative pain intensity will be assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain), both at rest and during movement.

SECONDARY OUTCOMES:
Total Postoperative Opioid Consumption | First 24 hours postoperatively
  Total opioid consumption during the first 24 hours postoperatively will be recorded using a patient-controlled analgesia (PCA) device and converted to morphine equivalent dose (mg).
Patient Satisfaction Score | Within the first 24 hours postoperatively
  Patient satisfaction with postoperative pain management will be assessed using a 5-point Likert Satisfaction Scale, ranging from 1 (very dissatisfied) to 5 (very satisfied), where higher scores indicate greater patient satisfaction.
Time to First Mobilization | Within the first 24 hours postoperatively
  Time to first mobilization after surgery will be recorded in hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Çam and Sakura City Hospital, Istanbul, BASAKSEHİR, Turkey (Türkiye)

REFERENCES:
- [Background] Roy R, Agarwal G, Pradhan C, Kuanar D. Total postoperative analgesia for hip surgeries, PENG block with LFCN block. Reg Anesth Pain Med. 2019 Mar 28:rapm-2019-100454. doi: 10.1136/rapm-2019-100454. Online ahead of print. No abstract available. PMID 30923252
- [Background] Yoo SH, Lee MJ, Beak MH, Kim WJ. Efficacy of Supplemental Ultrasound-Guided Pericapsular Nerve Group (PENG) Block Combined with Lateral Femoral Cutaneous Nerve Block in Patients Receiving Local Infiltration Analgesia after Hip Fracture Surgery: A Prospective Randomized Controlled Trial. Medicina (Kaunas). 2024 Feb 12;60(2):315. doi: 10.3390/medicina60020315. PMID 38399602
- [Background] Pascarella G, Costa F, Strumia A, Ruggiero A, Remore LM, Lanteri T, Hazboun A, Longo F, Gargano F, Schiavoni L, Mattei A, Agro FE, Carassiti M, Cataldo R. Lateral Femoral Cutaneous Nerve Block or Wound Infiltration Combined with Pericapsular Nerve Group (PENG) Block for Postoperative Analgesia following Total Hip Arthroplasty through Posterior Approach: A Randomized Controlled Trial. J Clin Med. 2024 May 2;13(9):2674. doi: 10.3390/jcm13092674. PMID 38731203
- [Background] Liang L, Zhang C, Dai W, He K. Comparison between pericapsular nerve group (PENG) block with lateral femoral cutaneous nerve block and supra-inguinal fascia iliaca compartment block (S-FICB) for total hip arthroplasty: a randomized controlled trial. J Anesth. 2023 Aug;37(4):503-510. doi: 10.1007/s00540-023-03192-6. Epub 2023 Apr 12. PMID 37043081